CLINICAL TRIAL: NCT04975191
Title: Personalized Feedback Programs for College Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HM20022611; R34AA027347 (NIH)
Record Dates: First submitted 2021-07-20; First posted 2021-07-23 (Actual); Results first posted 2023-05-31 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Alcohol Use, Unspecified
MeSH Terms: conditions — Alcohol Drinking | interventions — Health Resources; Body Mass Index

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Resources Program (RP) (Other)
  Interventions: Behavioral: Resources
- Personalized Feedback Program (PFP) (Active Comparator)
  Interventions: Behavioral: Personalized Feedback Program (PFP)
- Brief motivational intervention (BMI) (Active Comparator)
  Interventions: Behavioral: Substance Use Feedback Program (BMI)
- Combined PFP+BMI (Active Comparator)
  Interventions: Behavioral: Personalized Feedback Program (PFP); Behavioral: Substance Use Feedback Program (BMI)

INTERVENTIONS:
Behavioral: Resources — Participants will be provided a list of resources available at VCU that are intended to support student success
  Arms: Resources Program (RP)
Behavioral: Personalized Feedback Program (PFP) — Participants will complete an interactive online program that explores their personality-related traits to provide personalized recommendations for success
  Arms: Combined PFP+BMI; Personalized Feedback Program (PFP)
Behavioral: Substance Use Feedback Program (BMI) — Participants will complete an online program based on brief motivational intervention (BMI) content/principles that explores their current substance use patterns to make personalized recommendations for success
  Arms: Brief motivational intervention (BMI); Combined PFP+BMI

SUMMARY:
The purpose of this research study is to evaluate the effectiveness of different forms of personalized feedback intended to help students make their best personal choices to support their health and well-being in college.

DETAILED DESCRIPTION:
Risky substance use among college students is a widespread challenge that requires innovative prevention methods to address. A primary aim of this study is to assess the efficacy of receiving different types of personalized feedback on the substance use and wellbeing of college students. This preliminary efficacy will be evaluated through a multi-part randomized controlled trial comparing four conditions: (1) resources program, (2) on-line Personalized Feedback Program (PFP), (3) on-line Substance Use Feedback Program (based on brief motivational intervention (BMI) principles), and (4) PFP+BMI.

At the first time point, participants will be randomly selected into one of four conditions. Participants have an equal chance of being assigned to any one of the conditions. All participants will complete follow-up surveys at two additional timepoints (30 day follow-up; 3-month follow-up) to determine any changes that have occurred since they took part in their program at Time Point 1.

After the final survey, all participants, regardless of their initial group, will be invited to receive all of the personalized feedback components available across all conditions.

Findings from this study have great potential to enhance the effectiveness of college student substance use prevention programming and improve college student wellbeing.

ELIGIBILITY:
Inclusion Criteria:

* Consent: Voluntary consent must be provided.
* Age: Students over the age of 18 may participate.
* Year in college: Newly enrolled freshmen.
* Enrollment status: Only full-time VCU students will participate.

Exclusion Criteria:

* Age: Under the age of 18
* Year in College: A sophomore, junior or senior
* Enrollment Status: Enrolled part-time

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 252 (Actual)
Dates: Start 2021-08-29 (Actual); Primary Completion 2022-03-23 (Actual); Study Completion 2022-03-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Langberg, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Keyes, C. L. (2009). Brief description of the mental health continuum short form (MHC-SF). Scale retrieved from https://www.psytoolkit.org/survey-library/mhc-sf.html.
- [Result] Derogatis LR, Lipman RS, Covi L. SCL-90: an outpatient psychiatric rating scale--preliminary report. Psychopharmacol Bull. 1973 Jan;9(1):13-28. No abstract available. PMID 4682398
- [Result] Lamers SM, Westerhof GJ, Bohlmeijer ET, ten Klooster PM, Keyes CL. Evaluating the psychometric properties of the Mental Health Continuum-Short Form (MHC-SF). J Clin Psychol. 2011 Jan;67(1):99-110. doi: 10.1002/jclp.20741. PMID 20973032

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Resources Program (RP) | Personalized Feedback Program (PFP) | Brief Motivational Intervention (BMI) | Combined PFP+BMI
Started | 66 | 61 | 63 | 62
Completed | 52 | 56 | 53 | 52
Not Completed | 14 | 5 | 10 | 10
Not completed — Protocol Violation | 1 | 2 | 2 | 2
Not completed — Lost to Follow-up | 13 | 3 | 8 | 8

BASELINE CHARACTERISTICS:
Population: Not-completers lost to follow were included in baseline data analysis but not-completers due to protocol violations were not.
Groups:
- Total: Total of all reporting groups
Arm/Group | Resources Program (RP) | Personalized Feedback Program (PFP) | Brief Motivational Intervention (BMI) | Combined PFP+BMI | Total
Number analyzed (Participants) | 65 | 59 | 61 | 60 | 245
Age, Continuous [Mean (Standard Deviation); unit: years] | 18.28 (1.23) | 18.28 (0.57) | 18.26 (0.49) | 18.19 (0.41) | 18.25 (0.76)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex: Female | 57 | 41 | 54 | 48 | 200
  Sex: Male | 7 | 17 | 7 | 12 | 43
  Sex: Refuse to state | 1 | 1 | 0 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 4 | 0 | 0 | 4
  Asian | 14 | 16 | 11 | 6 | 47
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 1
  Black or African American | 12 | 9 | 10 | 10 | 41
  White | 33 | 23 | 28 | 29 | 113
  More than one race | 5 | 6 | 6 | 9 | 26
  Unknown or Not Reported | 0 | 1 | 6 | 6 | 13
Region of Enrollment [Number; unit: participants]
  United States | 65 | 59 | 61 | 60 | 245

OUTCOME MEASURES:

1. Primary Outcome: Change in Alcohol Use
Description: Number of participants who report alcohol use in the past 30 days
Time Frame: Baseline-3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Resources Program (RP) | Personalized Feedback Program (PFP) | Brief Motivational Intervention (BMI) | Combined PFP+BMI
Number analyzed (Participants) | 65 | 59 | 61 | 60
Participants | 19 | 17 | 22 | 18

2. Primary Outcome: Change in Cannabis Use
Description: Number of participants who report cannabis use in the past 30 days
Time Frame: Baseline-3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Resources Program (RP) | Personalized Feedback Program (PFP) | Brief Motivational Intervention (BMI) | Combined PFP+BMI
Number analyzed (Participants) | 65 | 59 | 61 | 60
Participants | 0 | 5 | 12 | 19

3. Secondary Outcome: Well-being as Assessed Using 14-item Questionnaire
Description: Well-being was measured with the 14 item Mental Health Continuum-Short Form (MHC-SF; Keyes, 2009; Lamers et al., 2011). Each item asks about past-month frequency of an aspect of positive mental health (e.g., I felt happy) with response options ranging from "never" to "every day." Higher scores reflect more positive well-being. Item scores ranged from 0 to 5 per item. Items were averaged to create a mean well-being measure for which measure scores ranged from a minimum of 0 to a maximum of 5.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Resources Program (RP) | Personalized Feedback Program (PFP) | Brief Motivational Intervention (BMI) | Combined PFP+BMI
Number analyzed (Participants) | 65 | 59 | 61 | 60
score on a scale | 2.91 (0.95) | 2.98 (0.99) | 2.98 (1.12) | 2.9 (1.07)

4. Secondary Outcome: Mental Health as Assessed Using 8-item Questionnaire
Description: Anxiety and depressive symptoms. Abbreviated scales from the Symptom Checklist-90 will be used to assess anxiety and depressive symptoms occurring within the last 30 days (Derogatis, Lipman, & Covi, 1973). Four items measured anxiety symptoms, and four items assessed depressive symptoms. Responses were rated on a 5-point Likert-type scale ("not at all", "a little bit", "moderately", "quite a bit", and "extremely"). Total scores were calculated for both the anxiety and depression subscales. The scores on each subscale ranged from a minimum of 0 to a maximum of 16. Higher scores reflect higher levels of anxiety and depression.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Resources Program (RP) | Personalized Feedback Program (PFP) | Brief Motivational Intervention (BMI) | Combined PFP+BMI
Number analyzed (Participants) | 65 | 59 | 61 | 60
score on a scale
  Anxiety | 5.12 (4.12) | 2.98 (3.42) | 4.00 (3.59) | 4.32 (4.35)
  Depression | 7.06 (3.68) | 6.46 (3.9) | 7.06 (4.35) | 7.09 (4.8)

5. Secondary Outcome: Resource Use
Description: Participants from each of the 4 groups were asked to indicate all of the VCU campus resources (e.g., recreation center, counseling center, writing center) they have utilized in the past 30 days from a list. Our team developed the list, which included 28 resources based on currently available resources for students at VCU. We summed the number of resources each participant used to create a "resource use score". Scores ranged from 0 to 28 and corresponded to the number of resources the participant reported using (e.g., if the participant reported using 3 of the resources on the list, they received a score of 3 on the scale). Higher values represent higher levels of resource use, that is, a better outcome. Mean scores for each group were calculated and are displayed on the outcomes table below.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: number of resources
Arm/Group | Resources Program (RP) | Personalized Feedback Program (PFP) | Brief Motivational Intervention (BMI) | Combined PFP+BMI
Number analyzed (Participants) | 65 | 59 | 61 | 60
number of resources | 2 (1.79) | 2.2 (2.23) | 1.52 (1.53) | 2.02 (2.09)

6. Secondary Outcome: Program Satisfaction
Description: Ten items are included to assess participants' opinions about their condition. Response options include "strongly disagree", "disagree", "neutral", "agree", and "strongly agree". Examples of the statements include "The length of the program was appropriate" and "I learned new information as part of this program." Total scores were averaged to create a mean satisfaction score. Mean scores ranged from a minimum of 0 to a maximum of 5. Higher scores represented higher satisfaction with the program whereas lower scores represented dissatisfaction with the program.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Resources Program (RP) | Personalized Feedback Program (PFP) | Brief Motivational Intervention (BMI) | Combined PFP+BMI
Number analyzed (Participants) | 65 | 59 | 61 | 60
score on a scale | 4.4 (3.68) | 3.83 (2.57) | 3.3 (3.38) | 4.3 (2.82)

7. Secondary Outcome: Risk Comprehension as Assessed Using 10-item Questionnaire
Description: Risk comprehension will be assessed using 10 questions related to participants' beliefs about what factors contribute to substance use and mental health. Correct responses for each question were scored as 1, and incorrect responses were scored as 0. Responses are summed to yield a single score. Scores ranged from a minimum of 0 to a maximum of 10. Higher scores indicate higher knowledge of risk for substance use problems.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Resources Program (RP) | Personalized Feedback Program (PFP) | Brief Motivational Intervention (BMI) | Combined PFP+BMI
Number analyzed (Participants) | 65 | 59 | 61 | 60
score on a scale | 8.33 (1.5) | 8.41 (1.78) | 8.53 (1.25) | 8.65 (1.42)

ADVERSE EVENTS:
Time Frame: NA - Adverse event data was not collected
Description: Adverse events data was not collected
Arm/Group | Resources Program (RP) | Personalized Feedback Program (PFP) | Brief Motivational Intervention (BMI) | Combined PFP+BMI
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2021-07-02): https://cdn.clinicaltrials.gov/large-docs/91/NCT04975191/Prot_001.pdf
  • Informed Consent Form (2021-10-18): https://cdn.clinicaltrials.gov/large-docs/91/NCT04975191/ICF_000.pdf